CLINICAL TRIAL: NCT01029379
Title: The Effect of Pharamocogenetices on Anesthesia Induction With Propofol
Brief Title: Pharmacogenetics of Propofol and Depth of Anesthesia
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Anna Oscarsson, Dr, University Hospital, Linkoeping
Other Study IDs: Progen1
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Anesthesia; Propofol
Keywords: propofol; depth of anesthesia; pharmacogenetics; Depth of anesthesia in correlation to plasma concentrations of propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 200 patients,ASA 1

SUMMARY:
Propofol, (2,6-diisopropylphenol) is a short-acting anesthetic drug used for induction and maintenance of anesthesia.

The aim of this study is to evaluate plasma concentrations of propofol in relation to depth of anesthesia, measured by continuous EEG and to correlate plasma concentrations with genetic analyses of liver enzymes responsible for drug elimination.

Our hypothesis is that there is an individual requirement of Propofol plasma concentration depending on genetic differences in drug elimination.

200 patients, ASA classification 1, planned for elective surgery of a duration of at least 30 minutes will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasian patents,
* (ASAclassification 1) planned for elective surgery,
* with body mass index 20-30,
* free from analgetic drug > 12 hours prior to anesthesia

Exclusion Criteria:

* Pregnancy,
* Smoking,
* allergy to propofol or peanuts,
* alcohol abuse,
* non-caucasian

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 200 patients, ASA classification 1 planned for elective surgery of at least 30 minutes duration
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
EEG pattern in correlation to clinical anesthesia | 20120101
  EEG pattern in correlation to clinical anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia and Intensive Care, Kalmar, Sweden

REFERENCES:
- [Derived] Khan MS, Zetterlund EL, Green H, Oscarsson A, Zackrisson AL, Svanborg E, Lindholm ML, Persson H, Eintrei C. Pharmacogenetics, plasma concentrations, clinical signs and EEG during propofol treatment. Basic Clin Pharmacol Toxicol. 2014 Dec;115(6):565-70. doi: 10.1111/bcpt.12277. Epub 2014 Jul 19. PMID 24891132